CLINICAL TRIAL: NCT05776927
Title: A Double-dummy, Double-blind, Randomized, Parallel-group, Active Controlled Study to Evaluate the Efficacy and Safety of QVM149 (Indacaterol Acetate / Glycopyrronium Bromide / Mometasone Furoate) Compared to Salmeterol Xinafoate/Fluticasone Propionate in Children From 12 Years to Less Than 18 Years of Age With Asthma.
Brief Title: A Study to Evaluate the Efficacy and Safety of QVM149 (Indacaterol Acetate / Glycopyrronium Bromide / Mometasone Furoate) Versus Salmeterol Xinafoate/Fluticasone Propionate in Children From 12 Years to Less Than 18 Years of Age With Asthma.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVM149C2301; 2022-502365-26 (Other: EU CTIS)
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Asthma; Adolescent; QVM149; Pediatric; LABA; LAMA; ICS; Triple Combination
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Fluticasone

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, parallel-group, active controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All site staff, including pharmacist will be blinded. All sponsor staff will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QVM149 (Experimental): QVM149 (Indacaterol as acetate 150 µg / glycopyrronium as bromide 50 µg / mometasone furoate 160 µg ) od delivered via Breezhaler® and Placebo to Salmeterol Xinafoate 50 μg
  / Fluticasone Propionate 500 μg bid delivered via Girohaler®
  Interventions: Drug: QVM149; Drug: Placebo to Salmeterol Xinafoate / Fluticasone Propionate; Drug: Run-In Medication; Drug: Rescue Medication; Device: Concept 1 Device; Device: Girohaler
- Salmeterol Xinafoate / Fluticasone Propionate Arm (Active Comparator): Salmeterol Xinafoate 50 μg / Fluticasone Propionate 500 μg bid delivered via Girohaler® and Placebo to QVM149 (Indacaterol as acetate 150 µg / glycopyrronium as bromide 50 µg / mometasone furoate 160 µg ) od delivered via Breezhaler®.
  Interventions: Drug: Salmeterol Xinafoate / Fluticasone Propionate; Drug: Placebo to QVM149; Drug: Run-In Medication; Drug: Rescue Medication; Device: Concept 1 Device; Device: Girohaler

INTERVENTIONS:
Drug: QVM149 — QVM149: Indacaterol as acetate 150 µg / glycopyrronium as bromide 50 µg / mometasone furoate 160 µg od delivered via Breezhaler®
  Arms: QVM149
Drug: Salmeterol Xinafoate / Fluticasone Propionate — Salmeterol Xinafoate 50 μg / Fluticasone Propionate 500 μg bid delivered via Girohaler®
  Arms: Salmeterol Xinafoate / Fluticasone Propionate Arm
Drug: Placebo to QVM149 — Placebo to QVM149: 150 μg Indacaterol Acetate / 50 μg Glycopyrronium Bromide / 160 μg Mometasone Furoate od delivered via Breezhaler®
  Arms: Salmeterol Xinafoate / Fluticasone Propionate Arm
Drug: Placebo to Salmeterol Xinafoate / Fluticasone Propionate — Placebo to Salmeterol Xinafoate 50 μg / Fluticasone Propionate 500 μg bid delivered via Girohaler®
  Arms: QVM149
Drug: Run-In Medication — Salmeterol Xinafoate 50 μg / Fluticasone Propionate 250μg bid delivered via Girohaler® or equivalent DPI device
Drug: Rescue Medication — Salbutamol 100μg / Albuterol 90μg
Device: Concept 1 Device — Concept1 (Breezhaler) used for QVM149 and placebo delivery
Device: Girohaler — Girohaler for Comparator and Placebo delivery.

SUMMARY:
A double-dummy, double-blind, randomized, parallel-group, active controlled study to evaluate the efficacy and safety of QVM149 (indacaterol acetate / glycopyrronium bromide / mometasone furoate) compared to salmeterol xinafoate/fluticasone propionate in children from 12 years to less than 18 years of age with asthma.

DETAILED DESCRIPTION:
This is a double-dummy, double-blind, randomized, parallel-group, 52 weeks, active controlled study to evaluate the efficacy and safety of indacaterol acetate 150 µg / glycopyrronium bromide 50 µg / mometasone furoate 160 µg (QVM149 150/50/160 µg) od in children from 12 to less than 18 years of age with asthma with pre-bronchodilator FEV1 ≥ 60 % and < 90 % of the predicted normal value for the participant.

The study duration of 60 weeks includes:

* a screening period of up to 15 days
* a run-in period of 14 days (run-in medication: salmeterol xinafoate/fluticasone propionate 50/250 µg bid)
* a treatment period of 52 weeks (either QVM149 150/50/160 µg od and placebo to salmeterol xinafoate/fluticasone propionate 50/500 µg bid, or salmeterol xinafoate/fluticasone propionate 50/500 µg bid and placebo to QVM149 150/50/160 µg od
* a safety follow up period of 30 days during which the participant will be back on standard of care treatment as appropriate.

ELIGIBILITY:
Inclusion criteria

Participants eligible for inclusion in this study must meet all of the following criteria:

1. Male and female adolescent subjects aged from equal to or greater than 12 years old to less than 18 years old at Screening visit.
2. Written and signed informed consent by parent(s)/legal guardian(s) for the pediatric participant and assent by the pediatric participant (depending on local requirements) must be obtained before any study-specific assessment is performed.
3. Patients with a documented diagnosis of persistent asthma (according to GINA 2022) for a period of at least 1 year prior to Screening.
4. Subjects who have used high dose ICS with LABA in combination for asthma for at least 3 months and at stable doses for at least 1 month prior to Screening.
5. Subjects must be symptomatic / inadequately controlled according to the investigator's opinion despite treatment with high stable doses of ICS with LABA in combination before Screening.
6. A history of one or more documented severe asthma exacerbations within the 12 months prior to Screening that required either:

   * Treatment with systemic corticosteroids (tablets, suspension or injection). OR
   * Hospitalization (defined as an in subject stay or greater than 24-hour stay in an observation area in the emergency room of other equivalent facility). NOTES: Investigators must use appropriate means to ensure the accuracy of the subject's exacerbation history (subject history at Screening documented in source notes, pharmacy records, hospital records, or chart records are acceptable).
7. Subjects must have ACQ-5 score equal to or greater than 1.5 at end of run-in visit prior to randomization (prior to double-blind treatment) and qualify for treatment with high dose LABA/ICS/LAMA.
8. Pre-bronchodilator FEV1 equal to or greater than 60 % and < 90 % of the predicted normal value for the subject according to ATS/ERS 2019 criteria after withholding bronchodilators (see Table 6-8) at both Run-in and before randomization.

   Withholding period of bronchodilators prior to spirometry:
   * SABA for equal to or greater than 6 hours
   * FDC or free combinations of ICS/LABA for equal to or greater than 48 hours
   * SAMA for equal to or greater than 8 hours
   * Xanthines equal to or greater than 7 days

   NOTES:
   * In case of combination ICS/LABA at screening, ICS alone should be continued until Run-in visit.
   * Wash-out period of each drug should be adhered to as above and should not be longer. If wash-out period is considered to be longer please contact the Novartis Medical Monitor.
   * A one-time repeat of percent predicted FEV1 (pre-bronchodilator FEV1) is allowed at Run-in as well as before randomization. Repeat of Run-in spirometry can be done later on the same day/visit (only to retest FEV1 criteria, not for reversibility, and before any salbutamol/albuterol inhalation) or in an ad-hoc visit to be scheduled on a later date (within 5 days of original Run-in) that would provide sufficient time to receive confirmation from the spirometry data central reviewer of the validity of the assessment before randomization. Run-in medication can be dispensed at Run-in but should be started only once the repeat spirometry was qualified by spirometry overread, if all inclusions at Run-in are successful in case of necessary repeat of Runin.
   * A one-time re-screen is allowed in case the subjects fail to meet the criteria at the repeat, provided the subjects return to their previous treatment until re-screening. In this circumstance, subjects are not required to go back on prior medication for 1 full month duration as outlined in inclusion criterion 4.
9. Subjects who demonstrate an increase in FEV1 of equal to or greater than 12% and 200 mL within 15 to 30 minutes after administration of 200-400 μg salbutamol/180-360 μg albuterol (or equivalent dose) at Run-in visit. All subjects must perform a reversibility test at Run-in visit that will be evaluated by central overread. If reversibility is not demonstrated at Run-in visit, or the assessment was evaluated as unacceptable by the central overread then:

   * Spirometry assessment to demonstrate Reversibility should be repeated once in an adhoc visit to be schedule preferably within 5 days. The reversibility test cannot be repeated on the same day because of the wash-out period of salbutamol/albuterol.
   * Subjects may be permitted to enter the study with historical evidence of reversibility that was performed according to ATS/ERS guidelines within 2 years prior to Screening.
   * Alternatively, subjects may be permitted to enter the study with a historical positive broncho-provocation test that was performed within 2 years prior to Screening. If reversibility is not demonstrated at Run-in visit (or after repeated assessment at ad-hoc visit within 5 days) with acceptable spirometry quality as per overread and historical evidence of reversibility/broncho-provocation is not available (or was not performed according to ATS/ERS guidelines) subjects must be screen failed and cannot be rescreened.

   Run-in medication can be dispensed at Run-in visit but should be started by the patient only if reversibility is met and all other elligibility criteria as per protocol are met.

   Spacer devices are permitted during reversibility testing only. The Investigator or delegate may decide whether to use spacer or not for the reversibility testing.
10. Subjects must meet all the following criteria at end of run-in visit prior to randomization:

    * Subjects must demonstrate acceptable inhaler devices (as per investigator judgement), peak flow meter, and spirometry techniques during the run-in period (from beginning to end of Run-in).
    * Subjects must demonstrate ≥ 70% compliance with the asthma controller ICS/LABA during the run-in period based on their inhaler use count. 70% compliance is defined as medication taken in 70% of the days in that period.
    * Subjects must demonstrate equal to or greater than 70% compliance with required use of the eDiary during the run-in period. 70% compliance is defined as completing the daily eDiary for 70% of the days (either morning or evening, including at least 7 morning and 7 evening eDiaries) during the Run-in period.

Exclusion criteria Participants meeting any of the following criteria are not eligible for inclusion in this study.

1. Subjects who have smoked or inhaled tobacco products within the 6 months period prior to Screening, or who have a smoking history of greater than 10 pack years (Note:1 pack is equivalent to 20 cigarettes. 10 pack years = 1 pack /day x 10 yrs., or ½ pack/day x 20 yrs.) or use of nicotine inhalers such as e-cigarettes at the time of Screening.
2. Subjects who have had an asthma attack/exacerbation requiring systemic steroids OR hospitalization (> 24 hours) OR emergency room visit (≤ 24 hours) within 6 weeks of Screening. If subjects experience an asthma attack/exacerbation requiring systemic steroids or emergency room visit between Screening and end of Run-in they may be rescreened 6 weeks after recovery from the exacerbation.
3. Subjects who have ever required intubation for a severe asthma attack/exacerbation.
4. Subjects who have a clinical condition which is likely to be worsened by ICS administration (e.g. glaucoma, cataract and fragility fractures) who are according to investigator's medical judgment at risk participating in the study.
5. Subjects who have had a respiratory tract infection or asthma worsening as determined by investigator within 4 weeks prior to Screening or between Screening and end of Run-in.

   Subjects may be re-screened 4 weeks after recovery from their respiratory tract infection or asthma worsening.
6. Subjects with evidence upon visual inspection (laboratory culture is not required) of clinically significant (in the opinion of investigator) oropharyngeal candidiasis at End of Run-in or earlier, with or without treatment. Subjects may be re-screened once their candidiasis has been treated and has resolved.
7. Subjects with any chronic conditions affecting the upper respiratory tract (eg. Chronic sinusitis) which in the opinion of the investigator may interfere with the study evaluation or optimal participation in the study.
8. Subjects with a history of chronic lung diseases other than asthma, including (but not limited to) sarcoidosis, interstitial lung disease, cystic fibrosis, clinically significant bronchiectasis and active tuberculosis.
9. Subjects with Type I diabetes or uncontrolled Type II diabetes.
10. Subjects who have a clinically significant laboratory abnormality as per investigator judgement or abnormal liver chemistry results (i.e. ALT, AST, total bilirubin, alkaline phosphatase, GGT and albumin above the upper limit of normal) before the end of run-in.
11. Use of other investigational drugs within 30 days or 5 half-lives of enrollment, or until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
12. Subjects who, either in the judgment of the investigator or the responsible Novartis personnel, have a clinically significant condition such as (but not limited to) unstable ischemic heart disease, New York Heart Association (NYHA) Class III/IV left ventricular failure arrhythmia, uncontrolled hypertension, cerebrovascular disease, psychiatric disease, neuro-degenerative diseases or other neurological diseases, uncontrolled hypoand hyper-thyroidism and other autoimmune diseases, hypokalemia, hyperadrenergic state, or ophthalmologic disorder or subjects with a medical condition that might compromise subject safety or compliance, interfere with evaluation, or preclude completion of the study. Subjects with paroxysmal (e.g., intermittent) atrial fibrillation are excluded. Subjects with persistent atrial fibrillation as defined by continuous atrial fibrillation for at least 6 months and controlled with a rate control strategy (i.e., selective beta blockers, calcium channel blocker, pacemaker placement, digoxin or ablation therapy) for at least 6 months may be considered for inclusion. In such subjects, atrial fibrillation must be present at the run-in visit with a resting ventricular rate < 100/min. At Run-In visit the atrial fibrillation must be confirmed by central reading.
13. Subjects with a history of myocardial infarction (this should be confirmed clinically by the investigator) within the previous 12 months.
14. Concomitant use of agents known to prolong the QTc interval unless it can be permanently discontinued for the duration of study.
15. Subjects with a history of long QT syndrome or whose QTc measured at Run-in or baseline prior to randomization (Fridericia method) is prolonged (> 450 msec for males and > 460 msec for females) and confirmed by a central assessor or inability to determine the QTcF interval (these subjects should not be re-screened).
16. Subjects who have a clinically significant ECG abnormality at Run-In visit and at any time during the Run-in period (including unscheduled ECG). ECG evidence of myocardial infarction at Run-in (via central reader) should be clinically assessed by the investigator with supportive documentation.
17. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
18. Subjects with a history of hypersensitivity or intolerance to any of the study drugs (including excipients) or to similar drugs within the class including untoward reactions to sympathomimetic amines or inhaled medication or any component thereof. This criteria also applies to rescue and Run-in medications.
19. Subjects who have not achieved an acceptable spirometry result at Run-in in accordance with American Thoracic Society/European Respiratory Society (ATS/ERS) criteria for acceptability and repeatability. Repeat spirometry may be allowed in an ad-hoc visit scheduled as close as possible from the first attempt (but not on the same day) if the spirometry did not qualify due to ATS/ERS criteria at Run-in. If the subjects fail the repeat assessment, the subjects may be re-screened once, provided the subjects return to their prior treatment until re-screened.
20. Subjects receiving any medications in the classes listed in Table 6-9.
21. Subjects receiving any asthma-related medications in the classes specified in Table 6-8 unless they undergo the required washout period and follow the adjustment to treatment program.
22. Subjects receiving medications in the classes listed in Table 6-10 should be excluded unless the medication has been stabilized for the specified period and the stated conditions have been met.
23. Subjects with severe narcolepsy and/or insomnia.
24. Subjects on Maintenance Immunotherapy (desensitization) for allergies for less than 3 months prior to Run-In or subjects on Maintenance Immunotherapy for more than 3 months prior to End of Run-In visit but expected to change throughout the course of the study.
25. Subjects who are serving a custodial sentence, do not have a permanent residence or who are detained under local mental health legislation/regulations.
26. Subjects who are directly associated with any members of the study team or their family members.
27. Subjects unable to use the Breezhaler® dry powder inhaler or the Girohaler® inhaler as per investigator 's judgement. Spacer devices are not permitted for rescue medication.
28. History of alcohol or other substance abuse.
29. Subjects with a known history of non-compliance to medication or who were unable or unwilling to complete a subject diary or who are unable or unwilling to use Electronic Peak Flow with e-diary device.
30. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test at Run-in.
31. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant (including female pediatric patients who are menarchal or who become menarchal during the study), unless they are using effective methods of contraception during dosing of study treatment. Effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps). For UK: with spermicidal foam/gel/film/cream/ vaginal suppository
    * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) In case of use of oral contraception females should have been stable on the same pill for a minimum of 3 months before taking investigational drug. The decision on the contraceptive method should be reviewed at least every 3 months to evaluate the individual need and compatibility of the method chosen.
32. Use of Long Acting Muscarinic Antagonist (LAMA) within 3 months prior to Screening.
33. History or presence of impaired renal function as indicated by clinically significant abnormal creatinine or blood urea nitrogen (BUN) and/or urea values, or abnormal urinary constituents (e.g. albuminuria) according to investigator's judgement.

    * Evidence of urinary obstruction, or difficulty in voiding
    * Evidence of congenital renal abnormalities with an established effect on renal function
    * Calculated eGFR <60 mL/min/1.73m2 using the Bedside Schwartz formula

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 304 (Estimated)
Dates: Start 2026-05-29 (Estimated); Primary Completion 2028-12-21 (Estimated); Study Completion 2029-12-24 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Trough FEV1 at Week 26. | Baseline, Week 26
  FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.

SECONDARY OUTCOMES:
Change from Baseline in Trough FEV1 at Week 52 | Baseline, Week 52
  FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
Change from Baseline in Asthma Control Questionnaire (ACQ-5) score at Week 26 and Week 52 | Baseline, Week 26, Week 52
  The ACQ-5 is a five-item, self-completed questionnaire, which is used as a measure of asthma control of a participant. The five questions (concerning nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheeze) enquire about the frequency and/or severity of symptoms over the previous week. The response options for all these questions range from zero (no impairment/limitation) to six (total impairment/ limitation) scale. ACQ-5 score range from 0 to 6. Higher scores indicates worsening of condition.
Change from Baseline in average Morning and Evening PEFR over 26 weeks and over 52 weeks treatment periods | Baseline, Week 26, Week 52
  Morning and Evening PEFR (Peak Expiratory Flow Rate) over 26 weeks and over 52 weeks
Change from Baseline in average Rescue medication use (daily, daytime, and nighttime) over 26 and 52 week treatment periods | Baseline, Week 26, Week 52
  Rescue medication use over 26 and 52 weeks treatment periods
Change from Baseline in Asthma Quality of Life Questionnaire (AQLQ(S)-12) total score at Week 26 and Week 52 | Baseline, Week 26, Week 52
  Asthma Quality of Life Questionnaire is a 32-item disease specific questionnaire designed to measure functional impairments that are most important to patients with asthma, with 7-point scale (1-totally limited/problems all the time, 7-not at all limited/no problems). It consists of 4 domains: symptoms, emotions, exposure to environmental stimuli and activity limitation. Mean score will be calculated for the four domains, as well as the overall quality-of-life score defined as the mean score of all 32 items.
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first dose up to 30 days after last dose (up to 56 weeks)
  Incidence of AEs and SAEs, including changes in vital signs, electrocardiograms (ECGs) and laboratory results qualifying and reported as AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.